CLINICAL TRIAL: NCT04537572
Title: A Comparison of Sample Collection Methods for SARS-COV-2 Antibody Testing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Salveo Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R2020-1002
Record Dates: First submitted 2020-09-01; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sample Collection Method (Other): All subjects will provide samples via traditional phlebotomy, finger-stick, and saliva collection.
  Interventions: Diagnostic Test: comparison of sample collection methods

INTERVENTIONS:
Diagnostic Test: comparison of sample collection methods — Samples will be collected via finger-stick, saliva collection, and traditional phlebotomy to determine effects on COVID-19 antibody test results.

SUMMARY:
The negative global consequences of the COVID-19 pandemic has prompted efforts to develop efficient laboratory testing protocols that can be quickly scaled in a practical way. Traditional phlebotomy requirements for antibody testing (venipuncture) often serve as a barrier to widespread population testing since they typically require dedicated facilities and personnel training. Conversely, antibodies are typically very stable in blood and require very little testing volume, which make antibody tests well suited to be run on samples collected via finger-stick, saliva, or other self-administered collection devices. Salveo Diagnostics is a CLIA/CAP certified clinical laboratory that routinely performs testing for anti-SARS-Cov-2 antibodies. The purposes of this protocol are to 1) assess the feasibility of streamlined sample collection procedures for assessing COVID-related immune status, and 2) to provide a mechanism for securing sequential samples in COVID positive and negative patients to support additional studies (e.g. investigating timing of anti-SARS-CoV-2 antibody class switching and antibody persistence).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed presence (N = 200) or absence (N = 100) of anti-SARS-COV2 antibodies
* >17 years old

Exclusion Criteria:

* Refusal or inability to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Laboratory determination of presence of anti-SARS-COV2 antibodies (IgM, IgA, and IgG) | testing will be performed within 2 days of collection

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Varvel, PhD, Principal Investigator — Salveo Diagnostics

IPD SHARING:
Plan to Share IPD: No